CLINICAL TRIAL: NCT00653536
Title: Feasibility and Safety of NeuroFlo™ in Patients With Persistent Arterial Occlusion (PAO) After Failed Mechanical Revascularization
Brief Title: A Study to Evaluate the Effects of the Neuroflo Device in People Who Have Had a Stroke
Acronym: PAO
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No Patients enrolled; sponsor not providing devices anymore
Sponsor: University of California, Los Angeles (Other)
Collaborators: CoAxia (Industry)
Responsible Party: Principal Investigator, David Liebeskind, Professor of Neurology, Associate Neurology Director, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-08-010
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Acute Stroke
Keywords: stroke; neuroflo; device; failure to recanalize
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: NeuroFlo — The device will be inflated for 45 minutes in acute ischemic stroke patients who have failed mechanical recanalization.

SUMMARY:
Patients with acute ischemic stroke and persistent arterial occlusion following failed mechanical revascularization, who can undergo NeuroFlo treatment within 18 hours of last time symptom free, will be eligible for enrollment to assess the safety and feasibility of the NeuroFlo catheter in treating ischemic stroke patients with persistent arterial occlusion following attempted thrombectomy. The NeuroFlo catheter is designed to partially obstruct the abdominal descending aorta thereby increasing blood flow to the brain. Cerebral perfusion is improved by diverting more blood through vessels as well as by expansion of the collateral circulation. Improved regional perfusion leads to clinical improvement.

DETAILED DESCRIPTION:
Patients with occlusion of a proximal artery experience prompt diversion of flow through collaterals and retrograde perfusion of the occluded arterial tree. Collateral perfusion sustains the penumbra and may lessen stroke severity provided recanalization of the occluded artery occurs. Thrombectomy attempts to achieve recanalization of the occluded artery, but 36% of patients (90/252 in MERCI and MultiMERCI studies) experienced persistent arterial occlusion (PAO, defined as TICI flow 0-1). PAO following attempted thrombectomy was associated with high mortality, with 53% dead at 90 days. Of the survivors, only 5% achieved mRS of 0-2. At present, there are no therapies that have been shown to improve these risks. Data obtained from a clinically indicated CT at 24 hours will be used to monitor for safety.

The safety endpoints for this study will be the proportion of patients who experience:

* Mortality and neurological deterioration (defined as an increase of ≥4 points on the NIHSS) at 5 days post treatment
* Change in neurological status and adverse events from baseline through 30 days from treatment

Other endpoints include:

* Change in neurological status and adverse events from baseline through 90 days from treatment
* The incidence of hemorrhagic transformation or other intracerebral bleeding will be assessed at 5 days post treatment.
* Cerebral blood flow changes associated with device therapy will be assessed through multimodal CT or MRI studies acquired at baseline and 3 hours post treatment.
* Potential patient benefit will be assessed through collection of neurological indices (NIHSS etc.) at baseline, 24 hours post-procedure, day 5 (or discharge), 30 days and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute cerebral ischemia due to occlusion of the internal carotid or middle cerebral artery
* NIHSS 8-25 (inclusive)
* Persistent arterial occlusion (defined as TICI 0 or 1) following failed mechanical revascularization (ref Table 2)
* Able to undergo NeuroFlo treatment within 18 hours of symptom onset (or from last time known normal)
* Informed consent from patient or legally authorized representative
* Negative pregnancy test in females of child-bearing potential

Exclusion Criteria:

* Etiology other than cerebral ischemia
* Acute hypodense parenchymal lesion or effacement of cerebral sulci in more than 1/3 of the middle cerebral artery territory
* Brainstem or cerebellar stroke
* Systolic blood pressure (BP) >220 mm Hg, or diastolic (BP) >140 mm Hg that cannot be lowered with medical management
* Any use of intravenous or intra-arterial thrombolytic medication
* Known secured or unsecured cerebral aneurysm or vascular malformation on CTA or MRA or history thereof
* Imaging evidence of current intracranial bleeding
* History of intracerebral hemorrhage
* Any aortic or femoral endovascular graft
* Aortic surgery within 6 weeks prior to the time of enrollment
* Known heparin sensitivity or allergy
* Participation in another therapeutic/treatment research protocol
* Any intracranial pathology interfering with the imaging assessments
* Current congestive or decompensated heart failure
* Known ejection fraction (EF) < 30% or evidence of NYHA Class IV or ACC/AHA Stage D heart failure within the past 3 months
* Known or echo evidence of aortic regurgitation ≥ 3+
* Myocardial infarction within last 3 months
* Evidence of acute MI on ECG or by cardiac enzymes
* Current or recent Class III or IV angina despite medical/surgical treatment
* INR > 1.7
* Platelet count < 100,000
* Creatinine > 1.5 times local laboratory standard
* Patients with cerebral arterial perforation or dissection due to attempted thrombectomy
* Patients with complications of femoral artery cannulation
* Patients with aortic diameter greater than 28 mm or smaller than 11 mm in diameter measured within 6 cm above and below the midpoint of the renal ostia (for 7Fr NeuroFlo Device)
* Evidence of aortic aneurysm
* High-grade iliac stenosis or vascular tortuosity that could prevent safe delivery and/or positioning of the NeuroFlo catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Mortality and neurological deterioration at 5 days post treatment | day 5

SECONDARY OUTCOMES:
Change in neurological status and adverse events from baseline through 30 days from treatment | Day 30
Change in neurological status and adverse events from baseline through 90 days from treatment | 90 days
Incidence of hemorrhagic transformation or other intracerebral bleeding at 5 days post treatment | day 5
Cerebral blood flow changes associated with device therapy assessed through multimodal MRI studies acquired at baseline and 3 hours post treatment obtained routinely at UCLA post IV or IA intervention in acute stroke patients | 3 hr and 24 hr

CONTACTS AND LOCATIONS:
Overall Officials: David S. Liebeskind, M.D., Principal Investigator — University of California, Los Angeles; Sidney Starkman, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States